CLINICAL TRIAL: NCT01382888
Title: Efficacy and Local Tolerability of Topically Applied Heparin (Heparin 2,400 IU /ml Cutaneous Spray) on the Suitability of Newly Constructed Primary Arteriovenous Fistulas in Patients Planned for Haemodialysis. A Multicentre, Randomized, Double-blind and Placebo-controlled Pilot Study
Brief Title: Efficacy and Local Tolerability of Topically Applied Heparin on the Suitability of Newly Constructed Primary Arteriovenous Fistulas in Patients Planned for Haemodialysis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor decided to terminate the study due to the low patient recruitment.
Sponsor: Cyathus Exquirere Pharmaforschungsgmbh (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CYT/Heparin - 01/11; 2011-000455-16 (EudraCT Number)
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Haemodialysis
Keywords: Haemodialysis; Arteriovenous fistula; Severe chronic kidney disease; Newly constructed primary arteriovenous fistulas in patients planned for haemodialysis
MeSH Terms: conditions — Arteriovenous Fistula; Renal Insufficiency, Chronic | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heparin 2,400 IU /ml Cutaneous Spray (Active Comparator): Patients are randomized to receive the active comparator heparin 2,400 IU/ml cutaneous spray for 24 weeks
  Interventions: Drug: Heparin 2,400 IU /ml Cutaneous Spray
- Placebo Cutaneous Spray (Placebo Comparator): Patients are randomized to receive placebo cutaneous spray for 24 weeks
  Interventions: Drug: Placebo Cutaneous Spray

INTERVENTIONS:
Drug: Heparin 2,400 IU /ml Cutaneous Spray — Randomization will be performed 2 - 14 days post fistula creation surgery following confirmation that the fistula is patent by physical examination. Patients that are randomized to this study arm, will be asked to administer the study medication twice daily. Patients will get adequate training before first administration.
  Arms: Heparin 2,400 IU /ml Cutaneous Spray
Drug: Placebo Cutaneous Spray — Randomization will be performed 2 - 14 days post fistula creation surgery following confirmation that the fistula is patent by physical examination. Patients that are randomized to this study arm, will be asked to administer the study medication (placebo) twice daily. Patients will get adequate training before first administration.
  Arms: Placebo Cutaneous Spray

SUMMARY:
The primary objective of this study is to evaluate the effect of topically applied heparin in comparison to placebo on suitability of newly constructed primary arteriovenous fistulas in patients planned for haemodialysis at 7th week (± 1 week) after first study drug administration.

DETAILED DESCRIPTION:
The clinical dilemma surrounding the maturation and suitability of the AVF in patients undergoing hemodialysis suggests the requirement for a medication that can be added to the standard therapy with in order to help maturation and suitability of newly created AVF. Numerous research papers published over the past 25 years indicate that heparin might have a positive impact on main factors involved in the early failure of native AVF to mature.

In total 56 eligible patients will be enrolled after giving informed consent. Screening will take place in the preceding 6 weeks before scheduled AVF creation. Only patients receiving a Brescia - Cimino (radio - cephalic) fistula or a distal ulnar artery to basilica vein, proximal radial artery to transposed basilica vein, brachial artery to transposed basilica vein and brachial artery to cephalic vein will later be randomized. Patients will be randomly assigned in equal proportions (each group 28 patients) to receive either topically applied heparin (Heparin 2,400 IU /ml Cutaneous Spray) or placebo using a computer-generated randomization. Participants and members of the study team will be blinded to treatment assignment. Patients will be instructed how to use and administer study medication for the consecutive 24 weeks following randomization.

Assessment of the primary endpoint (suitability of newly constructed primary arteriovenous fistulas) is done at 7th week (± 1 week) after first study drug administration. The suitability and unassisted patency and local safety and tolerability by physician and patient of the AVF will also be determined at 12 weeks (± 1 week) and 24 weeks (± 1 week) after first study drug administration. Administration of study medication will be stopped at week 24 after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female outpatients
* Aged over 18 years
* Stage 4 or 5 Chronic kidney Disease according to KDOQI classification
* Surgery to create an arteriovenous fistula in the lower arm is planned
* If female of childbearing potential: agree to maintain reliable birth control throughout the study and negative (urine) pregnancy test

Exclusion Criteria:

* Known hypersensitivity to any component of the study medication
* History of previous arm (side of planned AVF), neck, or chest surgery/trauma
* Anticipated kidney transplant from living donor within the next 3 months
* Presence of any comorbidity that limits patient's life expectancy to less than 6 months.
* Pregnancy / lactation or intention to fall pregnant during the time course of the study and women of childbearing potential who are not using adequate contraception
* Known bleeding disorder or established diagnosis of active or suspected bleeding
* Platelet count less than 80 x 10^9/L
* Uncontrolled hypertension: Diastolic blood pressure > 115 mm Hg or Systolic blood pressure > 200 mm Hg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Dialysis with a blood flow rate ≥ 300 ml/min OR, if the patient is not in need of dialysis, by combining the venous diameter > 0.4 cm and flow volume > 500ml/min assessed by duplex ultrasound, as well as via clinical impression | 7 ± 1 week
  Primary outcome measure is the suitability of the AVF (dialysis with a blood flow rate ≥ 300 ml/min ) at 7th week (± 1 week) after first study drug administration. Suitability of the AVF will be assessed by using the AVF for dialysis. If a flow rate of at least 300 ml/min can be reached for at least 3 minutes suitability is fulfilled.If the patient is not in need of dialysis, suitability will be assessed by combining the venous diameter > 0.4 cm and flow volume > 500ml/min assessed by duplex ultrasound, as well as via clinical impression

SECONDARY OUTCOMES:
Dialysis with a blood flow rate ≥ 300mL/min. If the patient is not in need of dialysis, by combining the venous diameter > 0.4 cm and flow volume > 500ml/min assessed by duplex ultrasound, as well as via clinical impression. | at 12th and 24th week after first study drug administration
  The suitability of the AVF (dialysis with a blood flow rate ≥ 300mL/min) at 12th and 24th week after first study drug administration. If a flow rate of at least 300 ml/min can be reached for at least 3 minutes suitability is fulfilled. If the patient is not in need of dialysis, the suitability will be assessed by combining the venous diameter > 0.4 cm and flow volume > 500ml/min assessed by duplex ultrasound, as well as via clinical impression.
The functional (unassisted) patency of AVF | at 7th, 12th and 24th weeks after first study drug administration
  Unassisted patency of the AVF will be assessed by palpation and auscultation for at least 30 seconds.
Local safety and tolerability profile of IMP by patients and investigator (Global assessment of tolerability) | 24 weeks
  A scale will be used to assess local tolerability. In addition the investigator will screen for known heparin specific reactions, i.e. skin rash and skin swelling.

CONTACTS AND LOCATIONS:
Locations (3):
- Austria (3):
  - Universitätsklinik für Innere Medizin III, Klinische Abteilung für Nephrologie und Dialyse, Medizinische Universität Wien, Vienna, Vienna
  - 6. Medizinische Abteilung mit Nephrologie und Dialyse, Wilhelminenspital Wien, Vienna, Vienna
  - Krankenhaus der Elisabethinen Linz, Linz